CLINICAL TRIAL: NCT02936986
Title: Endoscopic Ultrasound-guided Needle-based Confocal Laser Endomicroscopy for Diagnosis of Gastric Subepithelial Tumors
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Official Title: Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-21
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Gastric Subepithelial Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The differential diagnosis of gastric subepithelial tumors by endoscopic ultrasound is currently suboptimal. Needle-based confocal laser endomicroscopy (nCLE) is a novel endoscopic technique, which is compatible with the 19-gauge FNA needle. Under endoscopic ultrasonography (EUS) guidance, nCLE enables real-time in vivo imaging of lesion tissues at cellular and subcellular levels. This study aimed to describe nCLE interpretation criteria for the characterization of gastric subepithelial tumors, with histopathological correlation, and to perform the validation of these criteria.

ELIGIBILITY:
Derivative study

Inclusion Criteria:

* patients aged from 18 to 75 years, with gastric subepithelial tumors ≥ 2 cm

Exclusion Criteria:

* Previous EUS-FNA performed within the past 3 months, and usual contraindications to EUS-FNA, such as serous cardiopulmonary diseases, severe coagulopathy dysfunction, impaired kidney function
* Extramural structures, vascular lesions or cystic masses were visible by EUS
* Pregnancy or breastfeeding
* Known allergy to fluorescein sodium
* Inability to provide informed consent

Validation study

Inclusion Criteria:

* patients aged from 18 to 75 years, with gastric subepithelial tumors ≥ 1 cm

Exclusion Criteria:

* Previous EUS-FNA performed within the past 3 months, and usual contraindications to EUS-FNA, such as serous cardiopulmonary diseases, severe coagulopathy dysfunction, impaired kidney function
* Extramural structures, vascular lesions cystic masses or lipoma were visible by EUS
* Pregnancy or breastfeeding
* Known allergy to fluorescein sodium
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients undergoing EUS for the diagnosis of gastric subepithelial tumors will be recruited in this study at Qilu Hospital, Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The nCLE interpretation criteria for the characterization of gastric subepithelial tumors with histopathological correlation | 24 months
The feasibility, safety and diagnostic yield of nCLE for gastric subepithelial tumors | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Zhang MM, Zhong N, Wang X, Li CQ, Ji R, Li Z, Gu X, Yu YB, Li LX, Zuo XL, Li YQ. Endoscopic ultrasound-guided needle-based confocal laser endomicroscopy for diagnosis of gastric subepithelial tumors: a pilot study. Endoscopy. 2019 Jun;51(6):560-565. doi: 10.1055/a-0790-8436. Epub 2018 Dec 20. PMID 30572352